CLINICAL TRIAL: NCT00748280
Title: Pulpotomy Versus Root Canal Therapy to Treat Irreversible Pulpitis in Human Permanent Molars: A Multicenter Randomized Non-inferiority Trial.
Brief Title: Vital Pulp Therapy to Treat Irreversible Pulpitis
Acronym: VPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Saeed Asgary, Dean, Iranian Center foe Endodontic Research, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: C/B/4/8253
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Pulpitis
Keywords: Endodontics; CEM cement; Calcium enriched mixture; MTA; Root Canal Therapy; Pain; Pulpotomy; Human; Permanent; Molar teeth
MeSH Terms: conditions — Pulpitis; Pain | interventions — Pulpotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ORCT
  Interventions: Procedure: One-visit root canal therapy
- 2 (Experimental): PCEM/PMTA
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: One-visit root canal therapy — Teeth were isolated, caries was removed and access cavities were prepared. Canal preparation was conducted using step-back technique. The working lengths were determined and confirmed by radiographs. The minimum size file for preparing the working length was size ISO #25 K-file to within 0.5-2 mm of the radiographic apex of the root. During hand instrumentation, canals were frequently irrigated with adequate amount of sterile normal saline solution. The root canals were filled with multiple gutta-percha cones and sealer using lateral condensation technique. Placing a cotton pellet in the pulp chamber, the access cavity was temporarily filled. The treatments of all samples were performed one-visit.
  Other Names: single-visit RCT
  Arms: 1
Procedure: pulpotomy — Pulpotomy was performed with a large round bur in a high-speed handpiece with copious irrigation; removing inflamed pulp tissue to stump level. Hemostasis was achieved by irrigation of the cavity with sterile normal saline and application of small pieces of sterile cotton pellets. The blood clot-free pulpal wound was covered with approximately 2 mm layer of endodontic bio-materials, a sterile wet cotton pellet was then placed over the MTA/CEM cement and the cavity sealed with Cavit.
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of pulpotomy treatment (with new endodontic bio-materials) as a new treatment with one-visit root canal therapy as reference treatment in pain relief and clinical and radiographic success, for irreversible pulpitis of human permanent molar teeth.

DETAILED DESCRIPTION:
In one visit RCT (Arm 1): The teeth were anesthetized, isolated and endodontic access and instrumentation of all canals was done. Canal preparation was conducted using a step-back technique. The working lengths were determined and confirmed by radiography. Sterile normal saline solution was used for intra-canal irrigation. Root canals were obturated with gutta-percha and sealer using lateral condensation technique. After placing a cotton pellet in the pulp chamber, the access cavity was closed with Cavit.

In pulpotomy treatment with CEM/MTA (Arm 2): The teeth were anesthetized. Pulpotomy procedure of removing inflamed pulp tissue to the stump level was done. Homeostasis was achieved by irrigating the cavity with sterile normal saline and application of small pieces of sterile cotton pellets. The pulpal wound was covered with an approximately 2-mm-thick layer of MTA/CEM cement. Pulp chambers were then covered with a wet cotton pellet and sealed with Cavit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria:

  1. Patient reports pain of endodontic origin
  2. Diagnosis of irreversible pulpitis
* Eligibility criteria:

  1. Molar tooth
  2. Patient chooses to have tooth extraction for pain relief
  3. Age 9-65 years
  4. Both gender
  5. The patient had read and thoroughly understood the questionnaires; and
  6. Written informed consent
* Exclusion Criteria:

  1. Moderate or severe periodontitis
  2. None restorable tooth
  3. Internal or external root resorption
  4. Root canal calcification
  5. No bleeding after access cavity preparation
  6. Analgesic taken within the last 4 h
  7. Active systemic disease
  8. The patient was pregnant or nursing
  9. History of opioid addiction or abuse
  10. Temporary residency

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinical and radiographical success of pulpotomy with CEM cement | 5 year

SECONDARY OUTCOMES:
Patient Assessment of Pain - Visual Analogue Scale | 7 day

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jafar Eghbal, Prof., Study Director — Shahid Beheshti University of Medical Sciences; Jamileh Ghoddusi, Prof., Principal Investigator — Mashhad University of Medical Sciences
Locations (1):
- Iranian Center for Endodontic research, Tehran, Iran